CLINICAL TRIAL: NCT04057274
Title: Effect of a Single Bout of Moderate-intensity Aerobic Exercise on Colon Cancer Cell Growth in Vitro
Brief Title: Acute Effect of modeRate-intensity aerOBIc Exercise on Colon Cancer Cell Growth
Acronym: AEROBIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northumbria University (Other)
Collaborators: York St John University (Other); Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: AEROBIC2019
Record Dates: First submitted 2019-08-13; First posted 2019-08-15 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2019-09

CONDITIONS: Colon Adenocarcinoma; Colon Cancer
Keywords: Colon cancer; Aerobic exercise
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a randomised, counterbalanced, crossover study whereby all participants will complete an exercise assessment and a resting assessment in a randomised order.
Masking Description: It is not possible to blind participants nor investigators. Investigators will be blind to allocation order until after the first blood sample is drawn.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise assessment (Experimental): The exercise condition will involve venous blood samples being drawn immediately before and after a single bout of moderate-intensity aerobic interval exercise.
  Interventions: Other: Exercise assessment
- Resting assessment (No Intervention): The resting condition will involve venous blood samples being drawn before and after 60 minutes of seated rest.

INTERVENTIONS:
Other: Exercise assessment — The moderate-intensity aerobic interval exercise will be performed on a cycle ergometer under the supervision of trained staff in an exercise science laboratory. Participants will perform a 5 to 10-minute warm-up that begins by pedalling against a light resistance (60 W) and progressively increases in resistance until a target heart rate of 50-60% heart rate reserve is achieved. Participants will then complete 6 x 5-minute bouts at 60% heart rate reserve whilst maintaining a cadence of 60 rev·min-1, separated by 2.5-minutes of pedalling against light resistance (60 W). The session will finish with a cool-down at light resistance (60 W) lasting 10-minutes.
  Arms: Exercise assessment

SUMMARY:
This study involves drawing blood samples from men before and after they perform 30-minutes of moderate-intensity aerobic exercise. The investigators will evaluate whether adding the exercise serum to colon cancer cells in a dish can reduce the growth of the cells compared to the resting serum.

Note: serum is the liquid part of the blood that carries hormones and metabolites around the body.

DETAILED DESCRIPTION:
Regular exercise is associated with a reduced risk of developing colon cancer. However, the mechanisms underpinning the anti-cancer effect of exercise are not yet fully understood. A recent theory suggests that each time you exercise, the short-lasting spikes in circulating hormones can suppress the growth of cancer cells. Hence, every exercise bout could have a direct anti-cancer effect.

This study will recruit men with an increased of colon cancer and explore whether incubating colon cancer cells with serum collected after a bout of moderate-intensity aerobic exercise influences cell viability in vitro.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* BMI ≥ 25 kg/m2 and/or waist circumference of ≥ 94 cm
* Male
* Participating in less than 30 min of planned, structured, moderate to vigorous-intensity physical activity on three or more d·wk-1 for the last three months

Exclusion Criteria:

* Any absolute or relative contraindication to exercise testing, as determined by the American College of Sports Medicine
* Any sign/symptom of cardiovascular, metabolic or renal disease
* Known cardiovascular, metabolic or renal disease without written medical clearance from physician
* Resting hypertension (≥160 mmHg systolic and/or ≥90 mmHg diastolic)
* Chronic obstructive pulmonary disease and/or asthma with peak respiratory flow < 300 l/min
* Previous stroke or transient ischemic attack
* Epilepsy or aneurysm (large vessel or cerebral)
* Previous or current treatment for malignancy
* Clotting disorder
* Taking beta-adrenergic blocking agents
* Resting heart rate ≥ 100 bpm
* Musculoskeletal, neurological, anthropometric, or rheumatoid conditions that makes it not possible to pedal a bicycle and/or would be worsened due to exercise
* Body mass > 150 kg

Ages: 50 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Cell viability (%) | 48 hours
  Viability of a human colon cancer cell line (LoVo) will be assessed via quantification of the fluorescent signal by the resazurin assay (Sigma-Aldrich, Dorset, UK). Cells will be seeded in culture medium containing 10% serum from individual participants and incubated for 48 hours. Fluorescence will then be measured using a microplate reader at an excitation of 540 nm and emission of 590 nm. Background fluorescence will be subtracted from each well and then values will be normalised to fluorescence of control cells grown in 10% fetal bovine serum instead of participant serum to give a percent viability.

SECONDARY OUTCOMES:
Concentration of epinephrine (pg/ml) | Immediately before and immediately after the exercise and resting assessments
  Systemic concentration of epinephrine will be measured from serum
Concentration of norepinephrine (pg/ml) | Immediately before and immediately after the exercise and resting assessments
  Systemic concentration of norepinephrine will be measured from serum
Concentration of Interleukin 6 (pg/ml) | Immediately before and immediately after the exercise and resting assessments
  Systemic concentration of Interleukin 6 will be measured from serum
Concentration of Tumour Necrosis Factor alpha (pg/ml) | Immediately before and immediately after the exercise and resting assessments
  Systemic concentration of Tumour Necrosis Factor alpha will be measured from serum
Concentration of Insulin (pmol/l) | Immediately before and immediately after the exercise and resting assessments
  Systemic concentration of Insulin will be measured from serum
Concentration of Insulin-like growth factor 1 (ng/ml) | Immediately before and immediately after the exercise and resting assessments
  Systemic concentration of Insulin-like growth factor 1 will be measured from serum

CONTACTS AND LOCATIONS:
Overall Officials: Samuel T Orange, PhD, Principal Investigator — Northumbria University
Locations (2):
- United Kingdom (2):
  - York St John University Sports Park, York, North Yorkshire
  - Northumbria University City Campus, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Raw data and statistical code will be uploaded onto a publicly available repository
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Raw data will be made available immediately after publication of the aggregated data in a peer-reviewed Journal
Access Criteria: Publicly available

REFERENCES:
- [Background] Boyle T, Keegel T, Bull F, Heyworth J, Fritschi L. Physical activity and risks of proximal and distal colon cancers: a systematic review and meta-analysis. J Natl Cancer Inst. 2012 Oct 17;104(20):1548-61. doi: 10.1093/jnci/djs354. Epub 2012 Aug 22. PMID 22914790
- [Background] Dethlefsen C, Hansen LS, Lillelund C, Andersen C, Gehl J, Christensen JF, Pedersen BK, Hojman P. Exercise-Induced Catecholamines Activate the Hippo Tumor Suppressor Pathway to Reduce Risks of Breast Cancer Development. Cancer Res. 2017 Sep 15;77(18):4894-4904. doi: 10.1158/0008-5472.CAN-16-3125. PMID 28887324
- [Background] Dethlefsen C, Pedersen KS, Hojman P. Every exercise bout matters: linking systemic exercise responses to breast cancer control. Breast Cancer Res Treat. 2017 Apr;162(3):399-408. doi: 10.1007/s10549-017-4129-4. Epub 2017 Jan 30. PMID 28138894
- [Background] Devin JL, Hill MM, Mourtzakis M, Quadrilatero J, Jenkins DG, Skinner TL. Acute high intensity interval exercise reduces colon cancer cell growth. J Physiol. 2019 Apr;597(8):2177-2184. doi: 10.1113/JP277648. Epub 2019 Mar 20. PMID 30812059